CLINICAL TRIAL: NCT06841536
Title: Combined Effects of Statins and Exercise on Physiological Health Markers and Quality of Life in Patients With Dyslipidaemia
Brief Title: Combined Effects of Statins and Exercise on Training Sensitive Health Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Faroe Islands (Other)
Collaborators: University of Copenhagen (Other); Research council Faroe Islands (Unknown); National Hospital of the Faroe Islands (Other Government); Betri Stuðul (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0360; 2024-10 (Other: The Reasearch Ethics Board of the Faroe Islands)
Record Dates: First submitted 2025-02-08; First posted 2025-02-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia; Exercise training; Mitochondria; Aerobic capacity; Statins; Adaptation, Physiological; proteomics; genetics; quality of life
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin; Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized by block to achieve a 60 : 40 allocation between exercise and non-exercise conditions, stratified by (1) sex (male/female) and (2) prior statin use (yes/no). The four 12-week treatment arms are: 1) exercise + placebo, 2) exercise + atorvastatin (80 mg/day), 3) atorvastatin (80 mg/day) and 4) placebo for 12 weeks
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The above-mentioned are masked with regards to atorvastatin/placebo and not exercise/non-exercise
  Statistical analysis of primary outcome will be blinded to the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Atorvastatin + exercise (Active Comparator): Atorvastatin (80 mg) will be ingested once daily as oral tablets (80 mg/day). The starting dosage is 40 mg per day with a weekly increment of 40 mg reaching the maintenance dosage of 80 mg per day on week two. The titration protocol may be extended for participants with intolerable side-effects, and participants with intolerable side-effects at 80 mg may stay at a lower dosage (40 mg)
  Exercise: The exercise will be performed as supervised aerobic interval training sessions on cycling ergometers lasting ~45 min, four times weekly for 12 weeks. The exercise training will be conducted as a combination of high- and moderate-intensity interval training to ensure optimal adaptations of the primary outcomes.
  Interventions: Drug: Atorvastatin 80mg; Behavioral: Exercise
- Placebo + exercise (Other): Placebo (CaCO3) will be ingested once daily as oral tablets (volume-matched to atorvastatin group).
  Exercise: The exercise will be performed as supervised aerobic interval training sessions on cycling ergometers lasting ~45 min, four times weekly for 12 weeks. The exercise training will be conducted as a combination of high- and moderate-intensity interval training to ensure optimal adaptations of the primary outcomes.
  Interventions: Behavioral: Exercise
- Atorvastatin + non-exercise (Other): Atorvastatin (80 mg) will be ingested once daily as oral tablets (80 mg/day). The starting dosage is 40 mg per day with a weekly increment of 40 mg reaching the maintenance dosage of 80 mg per day on week two. The titration protocol may be extended for participants with intolerable side-effects, and participants with intolerable side-effects at 80 mg may stay at a lower dosage (40 mg)
  non-exercise: Participants are instructed to maintain habitual activity levels at the same level as when the participant was enrolled in the study.
  Interventions: Drug: Atorvastatin 80mg
- Placebo + non-exercise (No Intervention): Placebo (CaCO3) will be ingested once daily as oral tablets (volume-matched to atorvastatin group). Non-exercise: Participants are instructed to maintain habitual activity levels at the same level as when the participant was enrolled in the study.

INTERVENTIONS:
Drug: Atorvastatin 80mg — Daily intake of 80 mg of the approved drug Atorvastatin. Starting at dose 40 mg with 40 mg weekly increment reaching the maintenance dosage of 80 mg on week two, which is the approved maximum dosage of Atorvastatin. Participants who don't tolerate this fast up-titration may have prolonged tritation protocol (up to four weeks).
  Under special circumstances, participants with intolerable side-effects may stay at a lower dose (40 mg/day).
  The dosage and applied up-tritation is based on recommendations from trained cardiologists at the National Hospital of the Faroe Islands.
  Arms: Atorvastatin + exercise; Atorvastatin + non-exercise
Behavioral: Exercise — Exercise will be performed as aerobic interval training sessions on cycling ergometers lasting ~45 min, four times weekly for 12 weeks. All exercise sessions will be supervised. Participants will wear HR monitor system during all sessions (Polar Electro Oy, Kempele, Finland) and the Borg 6-to-20 scale will also be used to assess the rate of perceived exertion during exercise sessions. A 4-week ramp-up phase will be applied, consisting of two sessions in weeks 1 and 2, three sessions in weeks 3 and 4 after which participants will complete 4 sessions a week from weeks 5 to 12.
  Arms: Atorvastatin + exercise; Placebo + exercise

SUMMARY:
Around the world, about 4 in 10 adults have abnormal blood fat levels-known as dyslipidaemia-which raises their chances of getting heart disease. Many people with this condition are prescribed statins, medications that help lower the "bad" Low-density lipoprotein cholesterol (LDL-C) in the blood and, in doing so, help prevent serious heart-related problems. While statins do lower these harmful cholesterol levels, recent research suggests that statins might interfere with some of the positive effects that exercise typically has on muscle cells' energy centers (the mitochondria) and on a person's aerobic capacity. It is not yet fully understood how statins might influence these exercise benefits at the molecular level. To address this gap, the present study will look closely at how taking statins combined with a structured exercise program affects both the muscle cells and the whole-body fitness of people with dyslipidaemia. By using a wide-ranging protein analysis, the research aims to identify changes in muscle proteins and other metabolism-related factors that could explain why statins might alter the expected improvements from exercise.

Methods and Analysis In this 12-week study, we aim to enrol between 100 and 125 adults (aged 40-65 years, with dyslipidaemia without established heart disease); the trial is powered for the first 100, and recruitment will stay open up to 125 to offset potential drop-outs. Participants will be randomly split into one of four groups: (1) exercise plus a placebo (an inactive pill), (2) exercise plus a daily high-dose statin (atorvastatin, 80 mg), (3) a daily high-dose statin without exercise, or (4) a placebo without exercise. More participants will be placed in the exercise groups to better understand the combined effects of exercise and statins. The main measurement will be how well the muscle's mitochondria work, assessed by changes in an enzyme called citrate synthase (CS) from before the program to after. Other important measures will include overall fitness (using a peak oxygen uptake (VO2peak) test) and detailed protein analyses. The study will also look at genetic variations to see if they influence how each participant responds to the treatment.

Ethics and Sharing of Results The study has received approval from the Faroe Islands Ethical Committee (2024-10) and follows international guidelines to protect participants' rights and data. Once the research is complete, the findings will be shared in leading scientific journals for the broader public and medical community to learn from.

DETAILED DESCRIPTION:
Dyslipidaemia, defined by abnormal lipid profiles (including raised total cholesterol, LDL-C, and triglycerides, as well as reduced high-density lipoprotein cholesterol (HDL-C), affects close to 40% of adults aged 25 years and above worldwide. This condition significantly contributes to global morbidity and mortality. In particular, excess LDL-C has been associated with elevated atherosclerotic cardiovascular disease (ASCVD) risk due to its central role in cholesterol transport into the arterial wall, facilitating plaque formation and atherogenesis. The scale of the problem is illustrated by data indicating that high LDL-C levels were linked to approximately 4.40 million deaths and 98.62 million Disability-adjusted life years in 2019 alone. Notably, the highest regional prevalence of hypercholesterolaemia has been reported in Europe, where more than half of the adult population exhibits elevated plasma cholesterol concentrations. The reduction of circulating LDL-C, whether through pharmacological agents or lifestyle interventions, thus remains a key strategy in mitigating ASCVD risk.

Among available therapies, statins are a cornerstone of dyslipidaemia management due to their efficacy in lowering LDL-C and consequent reduction in cardiovascular event rates. For instance, decreasing LDL-C by 1 mmol/L through statin therapy is associated with up to a 20% reduction in both cardiovascular events and all-cause mortality. While pharmacotherapy is central to risk management, exercise training is also strongly recommended to improve lipid profiles and enhance cardiovascular health. Even relatively modest increases in cardiorespiratory fitness (CRF), on the order of approximately 1 metabolic equivalent (MET), translate into significant survival benefits of 10-25%. As cardiovascular diseases remain a leading global health concern, understanding how statins may interact with exercise-based interventions is essential for developing optimized treatment strategies for patients with dyslipidaemia.

Recent evidence suggests that the concurrent use of statins and structured exercise training does not always produce additive benefits, as initially presumed. In particular, some studies have reported that statin therapy may attenuate improvements in CRF and skeletal muscle mitochondrial function typically observed with endurance training. For example, administration of simvastatin at 40 mg/day hindered the usual exercise-induced increase in citrate synthase (CS) activity and aerobic capacity following 12 weeks of endurance exercise training in overweight adults. Similarly, high-dose atorvastatin (80 mg/day) has been shown to impair mitochondrial oxidative capacity in skeletal muscle, even in individuals free from overt cardiometabolic disease. These results are consistent with a growing body of work linking statin use to mitochondrial perturbations within skeletal muscle tissue. However, the precise biological mechanisms responsible for these observations remain poorly characterized. Modern omics approaches, such as untargeted proteomic profiling, may help elucidate how statins impact the network of mitochondrial proteins and metabolic pathways involved in exercise adaptation.

In addition to mitochondrial dysregulation, statin therapy-particularly at high doses-has been associated with a heightened risk of incident type 2 diabetes mellitus (T2DM). The underlying mechanisms appear multifactorial, involving alterations in insulin sensitivity and secretory function. Statins may diminish Glucose transporter type 4 (GLUT4)-mediated glucose uptake, affect mitochondrial energy transduction in skeletal muscle and adipose tissue, and promote lipotoxicity in pancreatic beta cells, collectively increasing insulin resistance and impairing normal insulin secretion. Thus, while statins robustly lower LDL-C and cardiovascular risk, their influence on glycemic control and metabolic health parameters warrants careful patient selection and ongoing glucose monitoring, especially in individuals predisposed to diabetes.

Musculoskeletal side effects, referred to as statin-associated muscle symptoms (SAMS), are another important consideration. Affecting an estimated 5-30% of statin users, SAMS range from mild myalgias to more significant muscle weakness, potentially prompting discontinuation of therapy and reducing adherence. This issue may also discourage regular physical activity and thereby negate some of the positive lifestyle modifications critical for long-term health management. Physical exertion may exacerbate these muscle symptoms, promoting a more sedentary pattern in individuals on statins. Although the pathophysiology of SAMS is not fully delineated, mitochondrial dysfunction related to impaired complexes III and IV activity, as well as reduced coenzyme Q10 availability, has been implicated.

Moreover, genetic polymorphisms can modulate statin pharmacodynamics and pharmacokinetics, potentially altering muscle tissue statin exposure and influencing inter-individual variability in both therapeutic and adverse responses to these agents. To date, however, the extent to which genetic variation might modify the interaction between statin therapy and exercise adaptations (on parameters such as mitochondrial function and systemic fitness) remains unknown.

In summary, although statins effectively diminish ASCVD risk by lowering LDL-C, emerging data suggest statins can reduce the beneficial effects of exercise training on skeletal muscle mitochondria and CRF. In addition, high-dose statin therapy may increase susceptibility to T2DM and aggravate muscle-related symptoms, thereby influencing the overall therapeutic benefit-risk profile. Despite considerable investigation in related areas, the precise molecular mechanisms underlying these effects, as well as the influence of genetics on this interplay, remain unclear. Notably, previous research has not yet encompassed a comprehensive, randomized, double-blinded, placebo-controlled trial that examines the simultaneous impact of statin therapy and structured exercise training on cardiovascular, muscular, and metabolic endpoints in dyslipidaemic individuals aged 40-65 years, including in-depth molecular phenotyping and genetic analyses.

Objective The present study aims to determine how statin therapy and exercise training, alone and in combination, influence whole-body aerobic capacity and mitochondrial function in individuals with dyslipidaemia but without established ASCVD. By employing untargeted proteomic methods, the investigation will identify molecular signatures and pathways through which statins may modify exercise-induced alterations in mitochondrial protein composition and metabolic phenotypes. An embedded sub-analysis will evaluate the role of genetic polymorphisms influencing statin pharmacodynamics and pharmacokinetics, thereby assessing how these genetic factors might shape individual variability in responses at both the muscle tissue and systemic levels. This integrative approach is expected to advance our understanding of the complex interactions between pharmacological lipid-lowering strategies and lifestyle interventions, ultimately guiding personalized management plans for patients with dyslipidaemia.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-65 years
* LDL-C > 4.0 mmol/L.

Exclusion Criteria:

* Diagnosed with serious chronic disease including type 1 or 2 diabetes.
* Cancer.
* A history of atherosclerotic cardiovascular disease.
* A history of major depression or other severe psychiatric disorders.
* Severe renal dysfunction (creatinine clearance <30 mL/min).
* Severe hepatic impairment.
* Active pregnancy or breast feeding.
* Active cigarette or e-cigarette smoker.
* Regular (>2 hours pr week) aerobic high-intensity exercise training.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Citrate synthase maximal activity (µmol/g/min) | Change from baseline to end-of-treatment (12 weeks)
  Maximal enzyme activity of citrate synthase will be determined from muscle homogenate using fluorometry

SECONDARY OUTCOMES:
Maximal oxygen uptake (ml/min) | Change from baseline to end-of-treatment (12 weeks)
  maximal oxygen uptake will be determined by a stepwise increased workload on a cycle ergometer
Targeted skeletal muscle proteomics | Change from baseline to end-of-treatment (12 weeks)
  Skeletal muscle proteomics targeted towards outcomes of interest related to oxidative/glycolytic pathway expression. Muscle samples will be analysed with data-independent parallel accumulation serial fragmentation (DIA-PASEF) mode on an Evosep One LC-system (Evosep, Denmark), in-line connected to a timsTOF SCP (Bruker). Data will be analysed in the DIA-NN software (v. 1.8.1) followed by bioinformatic analysis via RStudio
Lipid profile (mmol/L) | Change from baseline to end-of-treatment (12 weeks)
  Total cholesterol (mmol/L), low-density lipoprotein-cholesterol (mmol/L), high-density lipoprotein cholesterol (mmol/l) and triglycerides (mmol/l) will be measured from blood samples in a fasting state.
Concentration of lipoprotein (a) (nmol/L) | Change from baseline to end-of-treatment (12 weeks)
  Lipoprotein (a) will be measured from blood samples in a fasting state
Concentration of apolipoprotein B (nmol/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein B will be measured from blood samples in a fasting state
Statins (atorvastatin) accumulation in muscle tissue | Change from baseline to end-of-treatment (12 weeks)
  Measured from muscle tissue using ultrahigh-performance liquid chromatography-mass spectrometry (UHPLC-MS).
Skeletal muscle coenzyme Q10 | Change from baseline to end-of-treatment (12 weeks)
  Total coenzyme Q10 (CoQ10) content will be extracted from muscle tissue and quantified via an HPLC-ECD system
Body weight (kg) | Change from baseline to end-of-treatment (12 weeks)
  Weight will be measured to the nearest 0.1 kg. in a fasting state without shoes and wearing light clothes.
Fasting plasma glucose (mmol/L) | Change from baseline to end-of-treatment (12 weeks)
  Fasting plasma glucose will be measured from blood samples in a fasting state
Concentration of glycosylated hemoglobin A1c (HbA1c) (mmol/mol) | Change from baseline to end-of-treatment (12 weeks)
  HbA1c will be measured from blood samples in a fasting state
Blood pressure (mmHg) | Change from baseline to end-of-treatment (12 weeks)
  Systolic- and diastolic blood pressure will be measured in duplicate from the non-dominant arm with a digital blood pressure monitor in sitting position after at least 5 min of rest.
Resting heart rate (bpm) | Change from baseline to end-of-treatment (12 weeks)
  Resting heart rate will be measured in duplicate from the non-dominant arm with a digital blood pressure monitor in sitting position after at least 5 min of rest.
Steady-state systemic oxygen uptake (mL/min) | Change from baseline to end-of-treatment (12 weeks)
  steady-state systemic oxygen uptake (mL/min) is determined by indirect calorimetry during a submaximal cycle protocol on a cycling ergometer
Quality of life score | Change from baseline to end-of-treatment (12 weeks)
  The Short Form 36 Health Survey, which ranges from 0-100 for the overall domain scores with higher scores reflecting a higher quality of life.
Maximal 3-hydroxy-acetylCoa-dehydrogenase activity (µmol/g/min). | Change from baseline to end-of-treatment (12 weeks)
  Maximal enzyme activity of 3-hydroxy-acetylCoa-dehydrogenase activity will be determined from muscle homogenate using fluorometry
Maximal phosphofructokinase activity (µmol/g/min) | Change from baseline to end-of-treatment (12 weeks)
  Maximal phosphofructokinase activity will be determined from muscle homogenate using fluorometry
Waist and hip circumference (cm) | Change from baseline to end-of-treatment (12 weeks)
  Waist and hip circumference (cm) will be measured in duplicate after gentle expiration.
Body fat percentage (%) | Change from baseline to end-of-treatment (12 weeks)
  Whole-body fat percentage measured by bioelectrical impedance analysis (BIA) using the InBody 270 (InBody Co., Seoul, Korea).
Lean body mass (kg) | Change from baseline to end-of-treatment (12 weeks)
  Whole-body lean body mass measured by bioelectrical impedance analysis (BIA) using an InBody 270 device (InBody Co., Seoul, Korea).
Hand-grip strength (kg) | Change from baseline to end-of-treatment (12 weeks)
  maximal strength will be determined as voluntary maximal isometric contraction force of the non-dominant arm utilizing a JAMAR hand dynamometer
Mitochondrial expression of complex I (arbitrary units) | Change from baseline to end-of-treatment (12 weeks)
  Skeletal muscle mitochondrial biogenesis will be evaluated through expression of complex I using immunoblotting.
HOMA-IR | Change from baseline to end-of-treatment (12 weeks)
  Fasting Glucose [mg/dL] × Fasting Insulin [µU/mL]) / 405
Matsuda Index | Change from baseline to end-of-treatment (12 weeks)
  Calculated as 10,000/square root ([fasting glucose × fasting insulin × [mean glucose × mean insulin )])
Insulin secretion rate (ISR) | Change from baseline to end-of-treatment (12 weeks)
  Will be calculated from the OGTT
Oral disposition index | Change from baseline to end-of-treatment (12 weeks)
  Oral DI will be calculated as the product of oral insulin sensitivity index (ISI, same as Matsuda index) and oral insulin secretion index (ISR).
Statin-associated muscle symptoms (SAMS) | Change from baseline to end-of-treatment (12 weeks)
  Graded severity of muscle pain and/or tenderness (0-10) with higher scores reflecting worse SAMS.
Statin-associated muscle symptoms (SAMS) | Change from baseline to end-of-treatment (12 weeks)
  Graded severity of muscle tiredness and/or weakness (0-10) with higher scores reflecting worse SAMS.
Statin-associated muscle symptoms (SAMS) | Change from baseline to end-of-treatment (12 weeks)
  Graded severity of muscle complaints (0-10), with higher scores reflecting worse SAMS
Statin-associated muscle symptoms (SAMS) | Change from baseline to end-of-treatment (12 weeks)
  Muscle cramps (yes/no) and whether muscle complaint is symmetrical (yes/no)
Mitochondrial expression of complex II (arbitrary units) | Change from baseline to end-of-treatment (12 weeks)
  Skeletal muscle mitochondrial biogenesis will be evaluated through expression of complex II using immunoblotting.
Mitochondrial expression of complex III (arbitrary units) | Change from baseline to end-of-treatment (12 weeks)
  Skeletal muscle mitochondrial biogenesis will be evaluated through expression of complex III using immunoblotting.
Mitochondrial expression of complex IV (arbitrary units) | Change from baseline to end-of-treatment (12 weeks)
  Skeletal muscle mitochondrial biogenesis will be evaluated through expression of complex IV using immunoblotting.
Mitochondrial expression of complex V (arbitrary units) | Change from baseline to end-of-treatment (12 weeks)
  Skeletal muscle mitochondrial biogenesis will be evaluated through expression of complex V using immunoblotting.
Change in plasma Apolipoprotein A-I concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein A-I will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein A-II concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein A-II will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein A-IV concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein A-IV will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein B-100 concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein B-100 will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein B-48 concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein B-48 will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein C-II concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein C-II will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein C-III concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein C-III will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein D concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein D will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein E concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein E and its isoforms (He2, He4) will be measured from blood samples in a fasting state
Change in plasma Apolipoprotein H concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein H will be measured from blood samples in a fasting state
Change in plasma Clusterin (Apo J) concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Clusterin (Apo J) will be measured from blood samples in a fasting state
Apolipoprotein M concentration mg/dL (or g/L) | Change from baseline to end-of-treatment (12 weeks)
  Apolipoprotein M will be measured from blood samples in a fasting state
Change in plasma Cholesteryl Ester Transfer Protein (CETP) activity µmol cholesteryl-ester transferred · min-¹ · L-¹ (or "units /L") | Change from baseline to end-of-treatment (12 weeks)
  Cholesteryl Ester Transfer Protein (CETP) activity will be measured from blood samples in a fasting state
Change in plasma Lecithin-Cholesterol Acyltransferase (LCAT) activity nmol cholesteryl-ester formed · min-¹ · mL-¹ | Change from baseline to end-of-treatment (12 weeks)
  plasma Lecithin-Cholesterol Acyltransferase (LCAT) activity will be measured from blood samples in a fasting state
Change in plasma Albumin concentration (g/dL) | Change from baseline to end-of-treatment (12 weeks)
  plasma Albumin concentration will be measured from blood samples in a fasting state
Change in plasma Transthyretin concentration (mg/dL) | Change from baseline to end-of-treatment (12 weeks)
  plasma Transthyretin concentration will be measured from blood samples in a fasting state

OTHER OUTCOMES:
Anaerobic capacity | Change from baseline to end-of-treatment (12 weeks)
  Anaerobic capacity will be assessed by a 30-s Wingate Anaerobic test with a fixed resistance load in both men and women
Concentration of systemic coenzyme Q10 | Change from baseline to end-of-treatment (12 weeks)
  Measured from blood samples and using high-performance liquid chromatography (HPLC)
Total hemoglobin mass (g) | Change from baseline to end-of-treatment (12 weeks)
  Total hemoglobin mass (g) will be measured using the Carbon-monoxide rebreathing method.
Concentration of systemic markers of inflammation (fg/mL) | Change from baseline to end-of-treatment (12 weeks)
  Interferon gamma (fg/mL), tumor necrosis factor alpha (fg/mL) and interleukins 1beta, 2, 6, 8, 10 (fg/mL) as well as interleukin 1 receptor antagonist (IL-1ra) will be measured from blood sample
Concentration of C-reactive protein (mg/L) | Change from baseline to end-of-treatment (12 weeks)
  C-reactive protein will be measured from blood samples
Concentration of white blood cells (10^9/L) | Change from baseline to end-of-treatment (12 weeks)
  White blood cell count will be measured from blood samples
Telomere length | Change from baseline to end-of-treatment (12 weeks)
  Telomere length will be measured using quantitative polymerase chain reaction (qPCR).
Concentration of per- and polyfluoroalkyl substances (PFAS) | Change from baseline to end-of-treatment (12 weeks)
  PFAS concentrations will be measured in serum samples and using online-solid phase extraction and liquid chromatography coupled to a triple quadropole mass spectrometer (LC-MS/MS).
Rate of perceived exertion (RPE) during exercise sessions | Measured frequently throughout the intervention
  The Borg 6-to-20 scale where 6 means (no exertion) and 20 means (maximal exertion) will be used to assess the rate of perceived exertion following training sessions.
Rate of perceived exertion (RPE) during exercise capacity measurements | Change from baseline to end-of-treatment (12 weeks)
  The Borg 6-to-20 scale where 6 means (no exertion) and 20 means (maximal exertion) will be used to assess the rate of perceived exertion following sub-maximal and maximal exercise capacity.
Untargeted skeletal muscle proteomics | Change from baseline to end-of-treatment (12 weeks)
  Broader proteome coverage which may yield some interesting findings (explorative non-defined outcomes). Muscle samples will be analysed with data-independent parallel accumulation serial fragmentation (DIA-PASEF) mode on an Evosep One LC-system (Evosep, Denmark), in-line connected to a timsTOF SCP (Bruker). Data will be analysed in the DIA-NN software (v. 1.8.1) followed by bioinformatic analysis via RStudio

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Faroe Islands, Tórshavn, Faroe Islands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Kopin L, Lowenstein C. Dyslipidemia. Ann Intern Med. 2017 Dec 5;167(11):ITC81-ITC96. doi: 10.7326/AITC201712050. PMID 29204622
- [Background] Boren J, Chapman MJ, Krauss RM, Packard CJ, Bentzon JF, Binder CJ, Daemen MJ, Demer LL, Hegele RA, Nicholls SJ, Nordestgaard BG, Watts GF, Bruckert E, Fazio S, Ference BA, Graham I, Horton JD, Landmesser U, Laufs U, Masana L, Pasterkamp G, Raal FJ, Ray KK, Schunkert H, Taskinen MR, van de Sluis B, Wiklund O, Tokgozoglu L, Catapano AL, Ginsberg HN. Low-density lipoproteins cause atherosclerotic cardiovascular disease: pathophysiological, genetic, and therapeutic insights: a consensus statement from the European Atherosclerosis Society Consensus Panel. Eur Heart J. 2020 Jun 21;41(24):2313-2330. doi: 10.1093/eurheartj/ehz962. No abstract available. PMID 32052833
- [Background] Kokkinos PF, Faselis C, Myers J, Panagiotakos D, Doumas M. Interactive effects of fitness and statin treatment on mortality risk in veterans with dyslipidaemia: a cohort study. Lancet. 2013 Feb 2;381(9864):394-9. doi: 10.1016/S0140-6736(12)61426-3. Epub 2012 Nov 28. PMID 23199849
- [Background] Farrell SW, Finley CE, Grundy SM. Cardiorespiratory fitness, LDL cholesterol, and CHD mortality in men. Med Sci Sports Exerc. 2012 Nov;44(11):2132-7. doi: 10.1249/MSS.0b013e31826524be. PMID 22776869
- [Background] Mikus CR, Boyle LJ, Borengasser SJ, Oberlin DJ, Naples SP, Fletcher J, Meers GM, Ruebel M, Laughlin MH, Dellsperger KC, Fadel PJ, Thyfault JP. Simvastatin impairs exercise training adaptations. J Am Coll Cardiol. 2013 Aug 20;62(8):709-14. doi: 10.1016/j.jacc.2013.02.074. Epub 2013 Apr 10. PMID 23583255
- [Background] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Moreno-Cabanas A, Mora-Rodriguez R. Exercise Training Adaptations in Metabolic Syndrome Individuals on Chronic Statin Treatment. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz304. doi: 10.1210/clinem/dgz304. PMID 31875915
- [Background] Ryan TE, Torres MJ, Lin CT, Clark AH, Brophy PM, Smith CA, Smith CD, Morris EM, Thyfault JP, Neufer PD. High-dose atorvastatin therapy progressively decreases skeletal muscle mitochondrial respiratory capacity in humans. JCI Insight. 2024 Feb 22;9(4):e174125. doi: 10.1172/jci.insight.174125. PMID 38385748
- [Background] Allard NAE, Schirris TJJ, Verheggen RJ, Russel FGM, Rodenburg RJ, Smeitink JAM, Thompson PD, Hopman MTE, Timmers S. Statins Affect Skeletal Muscle Performance: Evidence for Disturbances in Energy Metabolism. J Clin Endocrinol Metab. 2018 Jan 1;103(1):75-84. doi: 10.1210/jc.2017-01561. PMID 29040646
- [Background] Paiva H, Thelen KM, Van Coster R, Smet J, De Paepe B, Mattila KM, Laakso J, Lehtimaki T, von Bergmann K, Lutjohann D, Laaksonen R. High-dose statins and skeletal muscle metabolism in humans: a randomized, controlled trial. Clin Pharmacol Ther. 2005 Jul;78(1):60-8. doi: 10.1016/j.clpt.2005.03.006. PMID 16003294
- [Background] Schirris TJ, Renkema GH, Ritschel T, Voermans NC, Bilos A, van Engelen BG, Brandt U, Koopman WJ, Beyrath JD, Rodenburg RJ, Willems PH, Smeitink JA, Russel FG. Statin-Induced Myopathy Is Associated with Mitochondrial Complex III Inhibition. Cell Metab. 2015 Sep 1;22(3):399-407. doi: 10.1016/j.cmet.2015.08.002. PMID 26331605
- [Background] Sirvent P, Bordenave S, Vermaelen M, Roels B, Vassort G, Mercier J, Raynaud E, Lacampagne A. Simvastatin induces impairment in skeletal muscle while heart is protected. Biochem Biophys Res Commun. 2005 Dec 23;338(3):1426-34. doi: 10.1016/j.bbrc.2005.10.108. Epub 2005 Oct 26. PMID 16271704
- [Background] Sirvent P, Mercier J, Vassort G, Lacampagne A. Simvastatin triggers mitochondria-induced Ca2+ signaling alteration in skeletal muscle. Biochem Biophys Res Commun. 2005 Apr 15;329(3):1067-75. doi: 10.1016/j.bbrc.2005.02.070. PMID 15752763
- [Background] Dirks AJ, Jones KM. Statin-induced apoptosis and skeletal myopathy. Am J Physiol Cell Physiol. 2006 Dec;291(6):C1208-12. doi: 10.1152/ajpcell.00226.2006. Epub 2006 Aug 2. PMID 16885396
- [Background] Muraki A, Miyashita K, Mitsuishi M, Tamaki M, Tanaka K, Itoh H. Coenzyme Q10 reverses mitochondrial dysfunction in atorvastatin-treated mice and increases exercise endurance. J Appl Physiol (1985). 2012 Aug;113(3):479-86. doi: 10.1152/japplphysiol.01362.2011. Epub 2012 May 31. PMID 22653988
- [Background] Bouitbir J, Charles AL, Rasseneur L, Dufour S, Piquard F, Geny B, Zoll J. Atorvastatin treatment reduces exercise capacities in rats: involvement of mitochondrial impairments and oxidative stress. J Appl Physiol (1985). 2011 Nov;111(5):1477-83. doi: 10.1152/japplphysiol.00107.2011. Epub 2011 Aug 18. PMID 21852406
- [Background] Kwak HB, Thalacker-Mercer A, Anderson EJ, Lin CT, Kane DA, Lee NS, Cortright RN, Bamman MM, Neufer PD. Simvastatin impairs ADP-stimulated respiration and increases mitochondrial oxidative stress in primary human skeletal myotubes. Free Radic Biol Med. 2012 Jan 1;52(1):198-207. doi: 10.1016/j.freeradbiomed.2011.10.449. Epub 2011 Oct 25. PMID 22080086
- [Background] Sirvent P, Fabre O, Bordenave S, Hillaire-Buys D, Raynaud De Mauverger E, Lacampagne A, Mercier J. Muscle mitochondrial metabolism and calcium signaling impairment in patients treated with statins. Toxicol Appl Pharmacol. 2012 Mar 1;259(2):263-8. doi: 10.1016/j.taap.2012.01.008. Epub 2012 Jan 17. PMID 22269104
- [Background] Schick BA, Laaksonen R, Frohlich JJ, Paiva H, Lehtimaki T, Humphries KH, Cote HC. Decreased skeletal muscle mitochondrial DNA in patients treated with high-dose simvastatin. Clin Pharmacol Ther. 2007 May;81(5):650-3. doi: 10.1038/sj.clpt.6100124. Epub 2007 Feb 28. PMID 17329991
- [Background] Meador BM, Huey KA. Statin-associated changes in skeletal muscle function and stress response after novel or accustomed exercise. Muscle Nerve. 2011 Dec;44(6):882-9. doi: 10.1002/mus.22236. PMID 22102458
- [Derived] Sjuretharson T, Larsen S, Jensen SBK, Bejder J, Rasmussen J, A Borg S, Kristiansen J, Meinhardsson JM, Olsen HW, Ellingsgaard H, Vigh-Larsen JF, Nordsborg NB, Mohr M. Investigating the combined effects of statins and exercise on skeletal muscle mitochondrial content and function, cardiorespiratory fitness and quality of life in individuals with dyslipidaemia: protocol for a randomised placebo-controlled trial. BMJ Open. 2025 Jun 5;15(6):e101425. doi: 10.1136/bmjopen-2025-101425. PMID 40473295

DOCUMENTS (1):
  • Statistical Analysis Plan (2026-01-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT06841536/SAP_001.pdf